CLINICAL TRIAL: NCT03405545
Title: High Intensity Interval Training and Skeletal Muscle Insulin Sensitivity: Unraveling Health Effects and Underlying Mechanisms
Brief Title: High Intensity Interval Training and Skeletal Muscle Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL62654.068.17
Record Dates: First submitted 2017-11-14; First posted 2018-01-23 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: 1 group of participants that performs 12 weeks of HIIT with metabolic measurements before and after this training period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIIT (Experimental): This group of subjects will perform High Intensity Interval training 3x/week for 12 weeks
  Interventions: Behavioral: High-intenstiy interval training

INTERVENTIONS:
Behavioral: High-intenstiy interval training — High-intensity interval training is a training of 30 minutes involving 10 bouts of 1 minute high intensity cycling (80-90% of maximum heart rate) interspersed by 2 minutes rest.

SUMMARY:
This human intervention study will test if 12 weeks of supervised HIIT-based intervention improves skeletal muscle NOGD capacity in obese subjects.

DETAILED DESCRIPTION:
19 overweight-obese (BMI => 27kg/m2), sedentary females and males aged 45-75yr will be enrolled in this study.

Participants will train 3 times/week under supervision during 12 weeks. Before, after and during this 12-week training period, there will be multiple metabolic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 45 - 75 years old
* Overweight to obese (BMI => 27kg/m2)
* Sedentary - subjects do not perform any regular physical activity weekly(<3 times per week, <150 min/week).

Exclusion Criteria:

* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Participation in an intensive weight-loss program or in vigorous exercise program during the last year before starting the study.
* HbA1c > 6.5% and glucose clearance rate >350 ml/kg/min (by OGTT).
* Previously diagnosed with type 2 diabetes
* Active cardiovascular disease. This will be determined by the questionnaires and by screening on medication.
* Use of beta-blockers
* Anticoagulant therapy
* Systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg
* Abuse of alcohol (> 3 units (1 unit = 10 gr ethanol) per day)
* Any contra-indication to Magnetic Resonance Imaging (MRI) scanning
* Participation in another biomedical study within 1 month before the first study visit, which may interfere with the outcomes of the present study.
* Use of any medication affecting the glucose homeostasis and whole body metabolism or diseases that may significantly interfere with the main aim of the study.
* Chronic renal dysfunction (creatinine >2 increased (normal value 64-104 µmol/l)
* Subjects who do not want to be informed about unexpected medical findings during the screening / study, or do not wish that their physician is informed, cannot participate in the study.
* Subjects will be included only when the dependent medical doctor of this study approves participation after evaluating all data obtained during the screening.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Non-oxidative glucose disposal | 9 hours
  Measured during a 2-step hyperinsulinemic-euglycemic clamp combined with indirect calorimetry

SECONDARY OUTCOMES:
Skeletal muscle glycogen content | 1 hour
  Assessed from skeletal muscle biopsies
Skeletal muscle insulin sensitivity | 9 hours
  Measured during a 2-step hyperinsulinemic-euglycemic clamp
24 hour glycaemic profile | 48 hours
  continuous glucose monitor
Skeletal muscle mitochondrial function assessed by Magnetic Resonance Spectroscopy Scan using 31P-MRS methodology, based on the phosphocreatine (PCr) recovery kinetics after exercise. | 1 hour
  The participant is positioned in the scanner with a home-built exercise device to perform consecutive knee-extensions, in which the participant has to lift a weight whilst laying in the scanner (50-60% max leg capacity of the subjects) for 5 minutes. Scout images of the upper leg are acquired and fine-tuned shimming is applied. Before, during and after exercise, spectra are acquired every 4 seconds. The restoration of PCr is driven almost purely by oxidative metabolism, the time to restore the normal amount reflects mitochondrial function (a faster restoration time means better mitochondrial function).
Metabolic Flexibility during exercise assessed by indirect calorimetry. | 30 minutes
  Participants will undergo a standardized cycling test at low, moderate and high intensity (30%-50%-70%) during 10 minutes each. Throughout the test, indirect calorimetry will be performed in order to measure changes in substrate oxidation during exercise.
Ectopic Fat accumulation in the liver assessed by magnetic resonance spectroscopy. | 1 hour
  Participants will undergo a magnetic resonance spectroscopy scan from which hepatic fat content will be quantified. In the 1H-MRS spectra, the water signal, that is dominating the proton spectra, will be suppressed using frequency-selective pre-pulse and the spectra will be fitted to quantify the lipid peak. A separate spectrum will be measured without water suppression to quantify the unsuppressed water signal. The CH2/Water ratio will be used as parameter of intrahepatic lipid content.
Maximal Acetylcarnitine formation in the upper-leg at rest and after exercise assessed by Magnetic Resonance Spectroscopy Scan | 1 hour
  Magnetic resonance imaging (MRI) will be used to guide the spectroscopy measurements and fine shimming will be performed to optimize the magnetic field homogeneity within the region of interest. A volume of interest will be selected within the m. vastus lateralis from the MRI images and the 1H-MRS spectra will be acquired from this region of interest. The intensity of the creatine signal will be used as internal reference.

OTHER OUTCOMES:
Effect of consumption of insulinogenic, CHO-rich drink post-exercise | 12 weeks
  Investigate whether the consumption of a insulinogenic, CHO-rich drink post-training prevention adverse effects related to blood glucose fluctuation while maintaining the effects of 12 weeks of HIIT on NOGD.

CONTACTS AND LOCATIONS:
Overall Officials: Matthijs Hesselink, Prof. PhD., Principal Investigator — Maastricht University; Vera Schrauwen-Hinderling, PhD, Principal Investigator — Maastricht University
Locations (1):
- University Maastricht, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No